CLINICAL TRIAL: NCT01714726
Title: A Phase 2a Study to Evaluate the Efficacy and Safety of MEDI2070 in Subjects With Moderate to Severe Crohn's Disease Who Have Failed or Are Intolerant to Anti-tumor Necrosis Factor-alpha Therapy
Brief Title: Evaluation of Efficacy and Safety of MEDI2070 in Patients With Active, Moderate-to-severe Crohn's Disease.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: MedImmune Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5170C00001; EudraCT number: 2012-004098-26; 2012-004098-26 (EudraCT Number)
Record Dates: First submitted 2012-10-24; First posted 2012-10-26 (Estimated); Results first posted 2019-03-06 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Crohn's Disease
Keywords: MEDI2070; inflammatory bowel disease; moderate to severe Crohn's disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — MEDI2070

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1 (Experimental): MEDI2070 iv infusion
  Interventions: Drug: MEDI2070
- 2 (Placebo Comparator): placebo iv infusion
  Interventions: Drug: placebo
- open-label (Experimental): MEDI2070 sc injection; open-label arm is available for all subjects upon completion of first placebo-controlled treatment period
  Interventions: Drug: MEDI2070

INTERVENTIONS:
Drug: MEDI2070 — 1 iv infusion on Week 0 and Week 4
  Arms: 1; open-label
Drug: placebo — 1 iv infusion on Week 0 and Week 4
  Arms: 2

SUMMARY:
The study is designed to evaluate the clinical efficacy and safety of MEDI2070 as compared to placebo. Investigational product will be administered as intravenous infusion in double-blind period, and as a subcutaneous injection in open-label period

DETAILED DESCRIPTION:
This is a two-part Phase 2a study compromising a 12-week, double-blind, placebo-controlled, treatment period followed by a 100-week, open label, treatment period to evaluate short-term efficacy, and the short- and long-term safety of MEDI2070 in subjects with moderate to severe, active CD who have failed or are intolerant to anti-TNFα therapy as determined by the investigator. Approximately 120 subjects will be randomized in a 1:1 ratio to initially receive a fixed IV dose of MEDI2070 or placebo on Week 0(Day1) and Week 4 (Day 29) during the 12-week, double-blind, placebo-controlled, treatment period. At the completion of the double-blind, placebo-controlled, treatment period (Week 12), subjects will have the option to enter a 100-week, open-label, treatment period where they will receive open-label MEDI2070 (SC) Q4W (Week 12 through Week 112). Subjects will be followed for safety at 3 visits over 28 weeks after their last dose of IP. Subjects will also be contacted by phone 36 weeks after their last dose of IP for safety.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed ileal, ileo-colonic, or colonic CD at least 6 months prior to screening.
* Men or women age 18 - 65 years at the time of screening.
* Moderate-sever active Crohn's Disease (CD), defined by a Crohn's Disease Activity Index (CDAI) score higher or equal 220 and lower or equal 450 at Day 1.
* No known history of active tuberculosis (TB).
* Received at least one anti-TNFα agent for the treatment of CD and did not initially respond.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Presence of ileostomy and/or colostomy.
* Short bowel syndrome.
* Bowel perforation or obstruction.
* History of cancer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2014-05-20 (Actual); Study Completion 2016-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (69):
- United States (25):
  - Research Site, Encinitas, California
  - Research Site, Los Angeles, California
  - Research Site, San Diego, California
  - Research Site, Torrance, California
  - Research Site, Lakewood, Colorado
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Macon, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Hammond, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Chevy Chase, Maryland
  - Research Site, Ann Arbor, Michigan
  - Research Site, Troy, Michigan
  - Research Site, Belton, Missouri
  - Research Site, New York, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Lima, Ohio
  - Research Site, Germantown, Tennessee
  - Research Site, San Antonio, Texas
  - Research Site, Seattle, Washington
- Canada (10):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Guelph, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Vaughan, Ontario
  - Research Site, Montreal, Quebec
- Czechia (5):
  - Research Site, České Budějovice
  - Research Site, Hradec Králové
  - Research Site, Litoměřice
  - Research Site, Ostrava-Poruba
  - Research Site, Prague
- France (5):
  - Research Site, Amiens
  - Research Site, Clichy
  - Research Site, Pessac
  - Research Site, Rouen
  - Research Site, Toulouse
- Germany (3):
  - Research Site, Hamburg
  - Research Site, München
  - Research Site, Potsdam
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Kaposvár
  - Research Site, Szombathely
- Italy (6):
  - Research Site, Bologna
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Roma
  - Research Site, Rozzano
- Poland (7):
  - Research Site, Bydgoszcz
  - Research Site, Opole
  - Research Site, Rzeszów
  - Research Site, Sopot
  - Research Site, Sosnowiec
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Spain (5):
  - Research Site, Barcelona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Sabadell(Barcelona)
  - Research Site, Seville
  - Research Site, Valencia

REFERENCES:
- [Background] Sands BE, Chen J, Feagan BG, Penney M, Rees WA, Danese S, Higgins PDR, Newbold P, Faggioni R, Patra K, Li J, Klekotka P, Morehouse C, Pulkstenis E, Drappa J, van der Merwe R, Gasser RA Jr. Efficacy and Safety of MEDI2070, an Antibody Against Interleukin 23, in Patients With Moderate to Severe Crohn's Disease: A Phase 2a Study. Gastroenterology. 2017 Jul;153(1):77-86.e6. doi: 10.1053/j.gastro.2017.03.049. Epub 2017 Apr 5. PMID 28390867
- [Derived] Danese S, Beaton A, Duncan EA, Mercier AK, Neisen J, Seth H, Zetterstrand S, Sands BE. Long-term safety of brazikumab in the open-label period of a randomized phase 2a study of patients with Crohn's disease. BMC Gastroenterol. 2023 Dec 20;23(1):451. doi: 10.1186/s12876-023-03078-7. PMID 38124112

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 174 screened subjects, 53 were considered screen failures. A total of 121 subjects were randomized, of which 2 did not receive study drug. Those 2 subjects were not included in the mITT population; therefore, those subjects are not counted in the participant flow.
Groups:
- Placebo: Participants received IV placebo concentrate and solvent for injection/infusion at week 0 and week 4.
- Experimental: MEDI2070 700mg: Participants received IV MEDI2070 700mg concentrate and solvent for injection/infusion at week 0 and week 4.
- Placebo/MEDI2070 210mg: Participants randomized to placebo arm in double-blind period received 210 mg SC MEDI2070 concentrate and solvent for solution injection/infusion every 4 week (Q4W) during the 100-week, open-label treatment period.
- MEDI2070 700mg/MEDI2070 210mg: Subjects randomized to MEDI2070 700mg arm in double-blind period received 210 mg SC MEDI2070 concentrate and solvent for solution for injection/infusion Q4W during the 100-week, open-label treatment period.
Period: Double-Blinded Induction Period
Arm/Group | Placebo | Experimental: MEDI2070 700mg | Placebo/MEDI2070 210mg | MEDI2070 700mg/MEDI2070 210mg
Started | 60 | 59 | 0 | 0
Completed | 52 | 52 | 0 | 0
Not Completed | 8 | 7 | 0 | 0
Not completed — Subject not in open label period | 3 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 3 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0
Period: Open-Label Period
Arm/Group | Placebo | Experimental: MEDI2070 700mg | Placebo/MEDI2070 210mg | MEDI2070 700mg/MEDI2070 210mg
Started | 0 | 0 | 52 | 52
Completed | 0 | 0 | 33 | 24
Not Completed | 0 | 0 | 19 | 28
Not completed — Other | 0 | 0 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 9 | 19
Not completed — Developed specific withdrawal criteria | 0 | 0 | 5 | 2
Not completed — Lost to Follow-up | 0 | 0 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Experimental: MEDI2070 700mg | Total
Number analyzed (Participants) | 60 | 59 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (10.7) | 34.8 (11.1) | 36.45 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 37 | 74
  Male | 23 | 22 | 45

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants With CDAI-70 Point Improvement at Week 8
Description: The CDAI is a multi-item instrument which measures severity of active Crohn's Disease monitored over 7 days and includes subject reported symptoms, physician-assessed signs, and laboratory markers. The CDAI score is calculated by summing weighted scores for subjective items (number of liquid or very soft stools, the degree of abdominal pain over a week and general well-being; and objective items (associated signs, use of anti-diarrhoeal medication, abdominal mass, haematocrit, daily morning temperature, and body weight). The CDAI scores range approximately from 0 to 600, with higher scores indicating greater disease activity. CDAI 70-point improvement is defined as a reduction from baseline in CDAI score of at least 70 points/scores, where baseline was the latest nonmissing observation prior to first administration of the study drug. Subjects in the mITT population were analysed for this end point.
Time Frame: Week 8
Population: Value of 0 represents the open-label portion of the trial
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Experimental: MEDI2070 700mg | Placebo/MEDI2070 210mg | MEDI2070 700mg/MEDI2070 210mg
Number analyzed (Participants) | 60 | 59 | 0 | 0
Percentage of Participants | 46.7 | 52.5 |  |

2. Secondary Outcome: Percentage of Participants With CDAI Response at Week 12
Description: The CDAI is a multi-item instrument which measures severity of active Crohn's Disease monitored over 7 days and includes subject reported symptoms, physician-assessed signs, and laboratory markers. The CDAI score is calculated by summing weighted scores for subjective items (number of liquid or very soft stools, the degree of abdominal pain over a week and general well-being; and objective items (associated signs, use of anti-diarrhoeal medication, abdominal mass, haematocrit, daily morning temperature, and body weight). The CDAI scores range approximately from 0 to 600, with higher scores indicating greater disease activity. CDAI response is defined by either a CDAI score of < 150 or a CDAI reduction from baseline of at least 100 points, where baseline was the latest non-missing observation prior to first administration of the study drug. Subjects in the mITT population were analysed for this end point.
Time Frame: Week 12
Population: Value of 0 represents the open-label portion of the trial
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Experimental: MEDI2070 700mg | Placebo/MEDI2070 210mg | MEDI2070 700mg/MEDI2070 210mg
Number analyzed (Participants) | 60 | 59 | 0 | 0
Percentage of Participants | 28.3 | 37.3 |  |

3. Primary Outcome: Percentage of Participants With Crohn's Disease Activity Index (CDAI) Response at Week 8
Description: A CDAI is a multi-item instrument which measures severity of active Crohn's Disease monitored over 7 days includes subject reported symptoms, physician-assessed signs, and laboratory markers. CDAI score = Sum of weighted scores for subjective items (number of liquid/soft stools, degree of abdominal pain, general well-being); and objective items (associated signs, use of anti-diarrhoeal medication, abdominal mass, haematocrit, daily morning temperature, body weight). CDAI scores range approximately from 0 to 600, higher scores indicating greater disease activity. The CDAI response at Week 8 is defined as either CDAI score of less than (<)150 or CDAI reduction from baseline of at least 100 points, where baseline was last non-missing observation prior to first administration of the study drug. Modified Intent-to-treat (mITT)population was analysed for this end point, which included all subjects who were randomized and received at least 1 dose of study drug in double-blind period.
Time Frame: Week 8
Population: Value of 0 represents the open-label portion of the trial
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Experimental: MEDI2070 700mg | Placebo/MEDI2070 210mg | MEDI2070 700mg/MEDI2070 210mg
Number analyzed (Participants) | 60 | 59 | 0 | 0
Percentage of Participants | 26.7 | 49.2 |  |
Statistical Analysis 1: Comparison: Placebo vs Experimental: MEDI2070 700mg; Test type: Superiority; p = 0.01, Regression, Logistic; Risk Difference (RD) = 22.5, 90% CI 2-sided [8.3 to 36.8]

4. Secondary Outcome: Percentage of Participants With CDAI Remission at Week 8
Description: The CDAI is a multi-item instrument which measures severity of active Crohn's Disease monitored over 7 days and includes subject reported symptoms, physician-assessed signs, and laboratory markers. The CDAI score is calculated by summing weighted scores for subjective items (number of liquid or very soft stools, the degree of abdominal pain over a week and general well-being; and objective items (associated signs, use of anti-diarrhoeal medication, abdominal mass, haematocrit, daily morning temperature, and body weight). The CDAI scores range approximately from 0 to 600, with higher scores indicating greater disease activity. The CDAI score of < 150 represent CDAI remission. Subjects in the mITT population were analysed for this end point.
Time Frame: Week 8
Population: Value of 0 represents the open-label portion of the trial
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Experimental: MEDI2070 700mg | Placebo/MEDI2070 210mg | MEDI2070 700mg/MEDI2070 210mg
Number analyzed (Participants) | 60 | 59 | 0 | 0
Percentage of Participants | 15 | 27.1 |  |

5. Secondary Outcome: Percentage of Participants With CDAI-100 Point Improvement at Week 8
Description: The CDAI is a multi-item instrument which measures severity of active Crohn's Disease monitored over 7 days and includes subject reported symptoms, physician-assessed signs, and laboratory markers. The CDAI score is calculated by summing weighted scores for subjective items (number of liquid or very soft stools, the degree of abdominal pain over a week and general well-being; and objective items (associated signs, use of anti-diarrhoeal medication, abdominal mass, haematocrit, daily morning temperature, and body weight). The CDAI scores range approximately from 0 to 600, with higher scores indicating greater disease activity. CDAI 100-point improvement is defined as a reduction from baseline in CDAI score of at least 100 points/scores, where baseline was the latest nonmissing observation prior to first administration of the study drug. Subjects in the mITT population were analysed for this end point.
Time Frame: Week 8
Population: Value of 0 represents the open-label portion of the trial
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Experimental: MEDI2070 700mg | Placebo/MEDI2070 210mg | MEDI2070 700mg/MEDI2070 210mg
Number analyzed (Participants) | 60 | 59 | 0 | 0
Percentage of Participants | 25.0 | 45.8 |  |

6. Secondary Outcome: Change From Baseline in CDAI Total Score at Week 8
Description: The CDAI is a multi-item instrument which measures severity of active Crohn's Disease monitored over 7 days and includes subject reported symptoms, physician-assessed signs, and laboratory markers. The CDAI score is calculated by summing weighted scores for subjective items (number of liquid or very soft stools, the degree of abdominal pain over a week and general well-being; and objective items (associated signs, use of anti-diarrhoeal medication, abdominal mass, haematocrit, daily morning temperature, and body weight). The CDAI scores range approximately from 0 to 600, with higher scores indicating greater disease activity. Subjects in the mITT population were analysed for this end point.
Time Frame: Week 8
Population: Value of 0 represents the open-label portion of the trial
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Experimental: MEDI2070 700mg | Placebo/MEDI2070 210mg | MEDI2070 700mg/MEDI2070 210mg
Number analyzed (Participants) | 60 | 59 | 0 | 0
Scores on a scale | -62.7 (13.5) | -99.0 (15.0) |  |

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) Double-blind Period
Description: An Adverse Event (AE) is any unfavourable and unintended sign, symptoms, or diseases temporally associated with use of study drug, whether or not considered related to study drug. A serious adverse event (SAE) is any AE that resulted in death, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, lifethreatening, a congenital anomaly/birth defect, or an important medical event. The TEAEs are defined as AEs present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug (Day 1) to 36 weeks post treatment (approximately 48 weeks). The safety population was analysed for this end point, which included all subjects who received any amount of study drug.
Time Frame: From study drug administration (Day 1) to 36 weeks post last blinded dose (up to 48 weeks)
Population: Value of 0 represents the open-label portion of the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Experimental: MEDI2070 700mg | Placebo/MEDI2070 210mg | MEDI2070 700mg/MEDI2070 210mg
Number analyzed (Participants) | 60 | 59 | 0 | 0
Participants | 41 | 40 |  |

8. Secondary Outcome: Number of Participants With Treatment Emergent Serious Adverse Events (TESAEs) in Double-blind Period
Description: as for outcome 7
Time Frame: From study drug administration (Day 1) to 36 weeks post last blinded dose (up to 48 weeks)
Population: Value of 0 represents the open-label portion of the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Experimental: MEDI2070 700mg | Placebo/MEDI2070 210mg | MEDI2070 700mg/MEDI2070 210mg
Number analyzed (Participants) | 60 | 59 | 0 | 0
Participants | 5 | 5 |  |

9. Secondary Outcome: Number of Participants With TEAEs in Open-label Period
Description: An AE is any unfavourable and unintended sign, symptoms, or diseases temporally associated with use of study drug, whether or not considered related to study drug. A SAE is any AE that resulted in death,inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, lifethreatening, a congenital anomaly/birth defect, or an important medical event. The TEAEs are defined as AEs present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug (Day 1) to 36 weeks post treatment (approximately 148 weeks). Open-label population was analysed for this endpoint, which included all subjects who were enrolled in the 100-week, open-label treatment period and have at least one dose of open-label MEDI2070 210 mg SC treatment.
Time Frame: From first open-label dose administration (Week 12) to 36 weeks post last dose (up to 148 weeks)
Population: Value of 0 represents the double-blind portion of the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Experimental: MEDI2070 700mg | Placebo/MEDI2070 210mg | MEDI2070 700mg/MEDI2070 210mg
Number analyzed (Participants) | 0 | 0 | 52 | 52
Participants |  |  | 44 | 43

10. Secondary Outcome: Number of Participants With TESAEs in Open-label Period
Description: as for outcome 9
Time Frame: From first open-label dose administration (Week 12) to 36 weeks post last dose (up to 148 weeks)
Population: Value of 0 represents the double-blind portion of the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Experimental: MEDI2070 700mg | Placebo/MEDI2070 210mg | MEDI2070 700mg/MEDI2070 210mg
Number analyzed (Participants) | 0 | 0 | 52 | 52
Participants |  |  | 8 | 12

11. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities as TEAEs in Double-blind Period
Description: The TEAEs are defined as AEs present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug (Day 1) to 36 weeks post treatment (up to approximately 48 weeks). Subjects in the safety population were analysed for this end point.
Time Frame: From study drug administration (Day 1) to 36 weeks post last blinded dose (up to 48 weeks)
Population: Value of 0 represents the open-label portion of the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Experimental: MEDI2070 700mg | Placebo/MEDI2070 210mg | MEDI2070 700mg/MEDI2070 210mg
Number analyzed (Participants) | 60 | 59 | 0 | 0
Participants
  Anaemia | 2 | 1 |  |
  Leukopenia | 0 | 1 |  |
  Neutropenia | 0 | 1 |  |
  Urine analysis Abnormal | 1 | 0 |  |
  Urine Abnormality | 0 | 1 |  |
  Urine bilirubin increased | 0 | 1 |  |
  Proteinuria | 0 | 1 |  |

12. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities Reported as TEAEs in Open-label Period
Description: The TEAEs are defined as AEs present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug (Day 1)to 36 weeks post treatment (up toapproximately 148 weeks). Open-label population was analysed for this endpoint, which included all subjects who were enrolled in the 100-week, open-label treatment period and have at least one dose of open-label MEDI2070 210 mg SC treatment.
Time Frame: From first open-label dose administration (Week 12) to 36 weeks post last dose (up to 148 weeks)
Population: Value of 0 represents the double-blind portion of the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Experimental: MEDI2070 700mg | Placebo/MEDI2070 210mg | MEDI2070 700mg/MEDI2070 210mg
Number analyzed (Participants) | 0 | 0 | 52 | 52
Participants
  Anaemia |  |  | 5 | 5
  Lymphocyte |  |  | 0 | 1
  Lymphopenia |  |  | 0 | 1
  Neutrophil count increased |  |  | 0 | 1
  Platelet count increased |  |  | 0 | 1
  Red cell distribution width increased |  |  | 0 | 1
  White blood cell count decreased |  |  | 0 | 1
  Chromaturia |  |  | 0 | 1
  Blood uric acid increased |  |  | 1 | 0
  Hypokalaemia |  |  | 1 | 1
  Hepatic enzyme increased |  |  | 0 | 1
  Hyperlipidemia |  |  | 1 | 0

13. Secondary Outcome: Number of Participants With Vital Signs Abnormalities Reported as TEAEs in Double-blind Period
Description: The TEAEs are defined as AEs present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug (Day 1)to 36 weeks post treatment(approximately 48 weeks). Subjects in the safety population were analysed for this end point.
Time Frame: From study drug administration (Day 1) to 36 weeks post last blinded dose (up to 48 weeks)
Population: Value of 0 represents the open-label portion of the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Experimental: MEDI2070 700mg | Placebo/MEDI2070 210mg | MEDI2070 700mg/MEDI2070 210mg
Number analyzed (Participants) | 60 | 59 | 0 | 0
Participants | 0 | 0 |  |

14. Secondary Outcome: Number of Participants With Vital Signs Abnormalities Reported as TEAEs in Open-label Period
Description: The TEAEs are defined as AEs present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug (Day 1) to 36 weeks post treatment(approximately 148 weeks). Open-label population was analysed for this endpoint, which included all subjects who were enrolled in the 100-week, open-label treatment period and have at least one dose of open-label MEDI2070 210 mg SC treatment.
Time Frame: From first open-label dose administration (Week 12) to 36 weeks post last dose (up to 148 weeks)
Population: Value of 0 represents the double-blind portion of the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Experimental: MEDI2070 700mg | Placebo/MEDI2070 210mg | MEDI2070 700mg/MEDI2070 210mg
Number analyzed (Participants) | 0 | 0 | 52 | 52
Participants |  |  | 0 | 0

15. Secondary Outcome: Maximum Mean Serum Concentration of MEDI2070 in Doubleblind Period
Description: Pharmacokinetic (PK) population included all subjects who received at least one dose of MEDI2070(either in double-blind period or in open-label period) and had at least one PK sample that was above the lower limit of quantification was considered for this end point. Serum concentration of MEDI2070 for subject in 'Placebo' arm is not applicable for this time frames and is reported by an arbitrary value (NA).
Time Frame: Post-dose on Week 0 (Day 1); pre and post-dose on Week 4; pre-dose on Week 8
Population: Serum MEDI2070 concentration data was summarized descriptively by visit. Value of 0 represents the open-label portion of the trial.
Measure: Mean (Standard Deviation); unit: mcg/ML
Arm/Group | Placebo | Experimental: MEDI2070 700mg | Placebo/MEDI2070 210mg | MEDI2070 700mg/MEDI2070 210mg
Number analyzed (Participants) | 60 | 59 | 0 | 0
mcg/ML
  Week 0 Post-dose (60, 58): number analyzed (Participants) | 60 | 58 | 0 | 0
  Week 0 Post-dose (60, 58) | NA (NA) — Serum concentration of MEDI2070 for subject in 'Placebo' arm is not applicable for this time frame | 186 (83.8) |  |
  Week 4 Pre-dose (54, 53): number analyzed (Participants) | 54 | 53 | 0 | 0
  Week 4 Pre-dose (54, 53) | NA (NA) — Serum concentration of MEDI2070 for subject in 'Placebo' arm is not applicable for this time frame | 37.4 (52.3) |  |
  Week 4 Post-dose (52, 51): number analyzed (Participants) | 52 | 51 | 0 | 0
  Week 4 Post-dose (52, 51) | NA (NA) — Serum concentration of MEDI2070 for subject in 'Placebo' arm is not applicable for this time frame | 209 (68.9) |  |
  Week 8 Pre-dose (55, 51): number analyzed (Participants) | 55 | 51 | 0 | 0
  Week 8 Pre-dose (55, 51) | NA (NA) — Serum concentration of MEDI2070 for subject in 'Placebo' arm is not applicable for this time frame | 39.2 (18.4) |  |

16. Secondary Outcome: Maximum Mean Serum Concentration of MEDI2070 in Open-label Period
Description: The PK population included all subjects who received at least one dose of MEDI2070 (either in double-blind period or in open-label period) and had at least one PK sample that was above the lower limit of quantification was considered for this end point. Serum concentration of MEDI2070 for subject in 'Placebo' arm is not applicable for pre-dose Week 12 time frame and is reported by an arbitrary value (NA).
Time Frame: Pre-dose on Weeks 12, 24, and 112
Population: Serum MEDI2070 concentration data was summarized descriptively by visit. Value of 0 represents the double-blind portion of the trial.
Measure: Mean (Standard Deviation); unit: mcg/ML
Arm/Group | Placebo | Experimental: MEDI2070 700mg | Placebo/MEDI2070 210mg | MEDI2070 700mg/MEDI2070 210mg
Number analyzed (Participants) | 0 | 0 | 52 | 52
mcg/ML
  Week 12 Pre-dose (51, 52): number analyzed (Participants) | 0 | 0 | 51 | 52
  Week 12 Pre-dose (51, 52) |  |  | NA (NA) — Serum concentration of MEDI2070 for subject in 'Placebo' arm is not applicable for this time frames | 16.7 (11.8)
  Week 24 Pre-dose (48, 43): number analyzed (Participants) | 0 | 0 | 48 | 43
  Week 24 Pre-dose (48, 43) |  |  | 14.5 (7.0) | 15.1 (6.38)
  Week 112 Pre-dose (24, 20): number analyzed (Participants) | 0 | 0 | 24 | 20
  Week 112 Pre-dose (24, 20) |  |  | 18.3 (7.73) | 22.4 (7.97)

17. Secondary Outcome: Number of Participants With Positive Anti-drug Antibody (ADA) to MEDI2070 in Double-blind Period
Description: The PK population included all subjects who received at least one dose of MEDI2070 (either in double-blind period or in open-label period) and had at least one PK sample that was above the lower limit of quantification was considered for this end point.
Time Frame: Baseline (Week0/Day 1) up to 28 week post last dose (approximately 40 weeks)
Population: Value of 0 represents the open-label portion of the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Experimental: MEDI2070 700mg | Placebo/MEDI2070 210mg | MEDI2070 700mg/MEDI2070 210mg
Number analyzed (Participants) | 60 | 59 | 0 | 0
Participants | 0 | 1 |  |

18. Secondary Outcome: Number of Participants With ADA Positive to MEDI2070 in Open-label Period
Description: as for outcome 17
Time Frame: Up to 28 week post last dose (approximately 140 weeks)
Population: Value of 0 represents the double-blind portion of the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Experimental: MEDI2070 700mg | Placebo/MEDI2070 210mg | MEDI2070 700mg/MEDI2070 210mg
Number analyzed (Participants) | 0 | 0 | 52 | 52
Participants |  |  | 1 | 1

ADVERSE EVENTS:
Time Frame: From study drug administration (Day 1) to 36 weeks post last dose (approximately 148 weeks)
Arm/Group | Placebo | Experimental: MEDI2070 700mg | Placebo/MEDI2070 210mg | MEDI2070 700mg/MEDI2070 210mg
Serious Adverse Events (participants affected / at risk) | 5/60 | 5/59 | 8/52 | 12/52
Other Adverse Events (participants affected / at risk) | 38/60 | 38/59 | 43/52 | 42/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=60) | Experimental: MEDI2070 700mg (N=59) | Placebo/MEDI2070 210mg (N=52) | MEDI2070 700mg/MEDI2070 210mg (N=52)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 12 (12)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=60) | Experimental: MEDI2070 700mg (N=59) | Placebo/MEDI2070 210mg (N=52) | MEDI2070 700mg/MEDI2070 210mg (N=52)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 5 (5) | 4 (4)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 4 (4) | 10 (10) | 12 (12) | 11 (11)
Pyrexia (General disorders) | 4 (4) | 1 (1) | 5 (5) | 3 (3)
Asthenia (General disorders) | 1 (1) | 2 (2) | 1 (1) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 6 (6) | 9 (9) | 10 (10)
Crohn's disease (Gastrointestinal disorders) | 3 (3) | 3 (3) | 6 (6) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 7 (7) | 7 (7)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 5 (5) | 6 (6)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3) | 8 (8) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 5 (5)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 5 (5) | 5 (5)
Nasopharyngitis (Infections and infestations) | 6 (6) | 9 (9) | 8 (8) | 15 (15)
Sinusitis (Infections and infestations) | 4 (4) | 0 (0) | 3 (3) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 5 (5) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 8 (8) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 8 (8) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 5 (5) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 4 (4)

LIMITATIONS AND CAVEATS:
A formal statistical analysis was not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo. (Note that this agreement language may appear in the study protocol)